CLINICAL TRIAL: NCT06714812
Title: Characteristics of Diarrheal Adverse Events in a Caucasian Population of Patients With Idiopathic Pulmonary Fibrosis Undergoing Treatment With Nintedanib - Pilot Study
Brief Title: Diarrheal Adverse Events in Caucasian Patients With Idiopathic Pulmonary Fibrosis Undergoing Treatment With Nintedanib
Acronym: EAD-IPF-N
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: EAD-IPF-N
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: IPF
Keywords: IPF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to identify the demographic and clinical characteristics associated with the development of diarrheal adverse events in a Caucasian population with IPF undergoing treatment with nintedanib. Additionally this study aims to evaluate the different therapeutic strategies for dose reduction of nintedanib and assess the effectiveness of these strategies in reducing the occurrence of diarrhea.

DETAILED DESCRIPTION:
The study population consists of patients treated with Nintedanib for IPF who are followed at the Interstitial Lung Disease Outpatient Clinic of the Pneumology and Respiratory Intensive Care Unit at the IRCCS Azienda Ospedaliero-Universitaria of Bologna, Policlinico di Sant'Orsola, and who have received the treatment for at least 12 consecutive months.

At the first available visit (which will be conducted according to the routine follow-up schedule), informed consent for partecipation in the study will be obtained. Following the signing of the informed consent, the data relevant to the protocol will be collected retrospectively, concerning the visit at which nintedanib therapy was initiated and the follow-up visits conducted at 6 and 12 months from the start of the antifibrotic therapy, as per clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian ethnicity;
* Age ≥ 18 years;
* Subjects with a diagnosis of IPF who started antifibrotic therapy with nintedanib on or after 01/06/2020.
* Obtaining written informed consent

Exclusion Criteria:

* clinical and functional data not availbale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Nintedanib for IPF who are seen at the Interstitial Lung Disease Outpatient Clinic of the Pneumology and Respiratory Intensive Care Unit at the IRCCS Azienda Ospedaliero-Universitaria of Bologna, Policlinico di Sant'Orsola, and who have received the treatment for at least 12 consecutive months.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of the demographic and clinical characteristics associated with the development of diarrheal adverse events in a Caucasian population with IPF undergoing treatment with nintedanib | 18 months
  Presence and intensity of diarrheal adverse events defined according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, which defines diarrhea as 'frequent and watery bowel movements' and classifies it into the following grades:
  Grade 1 = Increase in the number of daily bowel movements < 4 compared to baseline.
  Grade 2 = Increase in the number of daily bowel movements from 4-6 compared to baseline.
  Grade 3 = Increase in the number of daily bowel movements > 7 compared to baseline.
  Grade 4 = Requires urgent intervention, life-threatening. Grade 5 = Death

SECONDARY OUTCOMES:
Identification of the functional parameters associated with the temporary dose reduction of nintedanib | 18 months
  Temporary dose reduction of nintedanib
Evaluation of the proportion of patients requiring a permanent dose reduction of nintedanib (100 mg twice daily) or discontinuation of the drug, and comparison of their characteristics with those patients who did not require therapy modifications. | 18 months
  Permanent reduction or discontinuation of nintedanib. Dose reduction of nintedanib is defined as the transition from the 'full' dose-equivalent to taking one 150 mg capsule twice daily-to the 'reduced' dose-equivalent to taking one 100 mg capsule twice daily. 'Reduction' and 'discontinuation' of nintedanib are considered two distinct outcomes.
Assessment of the effectiveness of different nintedanib dose reduction strategies in reducing diarrheal symptoms | 18 months
  Effectiveness of the dose reduction strategy, defined as a decrease of at least 1 grade on the CTCAE scale.
Calculation of the incidence of diarrheal adverse events in a Caucasian population of patients with IPF undergoing antifibrotic treatment with nintedanib during the first year of therapy | 18 months
  Number of diarrheal adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nava, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliera-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided